CLINICAL TRIAL: NCT01353742
Title: A Randomized, Open-label, Single-dose, Two-period, Crossover Study to Demonstrate the Bioequivalence of the Fixed Dose Combination (FDC) of Lamivudine and Adefovir Dipivoxil (100mg/10mg) to Heptodin® (100mg ) and Hepsera® (10mg)
Brief Title: Lamivudine and Adefovir Dipivoxil Fixed Dose Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114957
Record Dates: First submitted 2011-05-05; First posted 2011-05-16 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamivudine and Adefovir dipivoxil (Active Comparator): One 100mg Lamivudine tablet and One 10mg Adefovir dipivoxil tablet
  Interventions: Drug: Lamivudine; Drug: Adefovir dipivoxil
- Fixed dose combination (Experimental): One capsule (100mg lamivudine and 10mg adefovir dipivoxil)
  Interventions: Drug: Fixed dose combination (Lamivudine and Adefovir dipivoxil)

INTERVENTIONS:
Drug: Lamivudine — 100mg tablet
  Other Names: Heptodin
  Arms: Lamivudine and Adefovir dipivoxil
Drug: Adefovir dipivoxil — 10mg tablet
  Other Names: Hepsera
  Arms: Lamivudine and Adefovir dipivoxil
Drug: Fixed dose combination (Lamivudine and Adefovir dipivoxil) — 100mg/10mg capsule
  Other Names: FDC
  Arms: Fixed dose combination

SUMMARY:
This is a phase I study being conducted to support the clinical development program of a FDC product of the nucleoside analogue lamivudine and the nucleotide analogue adefovir dipivoxil. To establish bioequivalence, the exposure of lamivudine and adefovir dipivoxil when administered as the FDC will be compared to that of Heptodin (lamivudine) and Hepsera (adefovir dipivoxil) when administered separately. In this study, the FDC product will contain 100mg lamivudine/10mg adefovir dipivoxil.

Total 40 healthy adult subjects will be enrolled. The study will include a screening visit and two treatment sessions. The screening visit will be conducted up to 3 weeks prior to the first dose of Session 1. All subjects will receive Regimen A through B according to the randomization schedule. Eligible subjects will be enrolled in the study and randomized to receive the following treatment regimens in table below in one of the following treatment sequences: AB, or BA. There will be a seven to ten days washout period between each treatment session. Pharmacokinetic sampling for measurement of plasma lamivudine and adefovir dipivoxil concentrations will be conducted over a 48-hour period following the morning administration of study medication in each study session. During this time, all subjects will remain in the unit for pharmacokinetic (PK) sample collection. The total duration (from screening to the end of the study) of each subject's participation will be approximately four weeks.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) infection is common, with an estimated global prevalence of more than 400 million people, or approximately 5% of the world's population. Chronic hepatitis B virus (HBV) carriers with evidence of ongoing viral replication are at highest risk for the development of active liver inflammation (i.e., hepatitis B) and progressive liver disease. They are also the major contributor to the spread of HBV infection.

The goals of therapy in CHB include suppression of HBV replication, reduction of necroinflammatory processes in the liver, and prevention of progression to serious liver disease or death. The HBV polymerase has an error rate that is intermediate between that of human immunodeficiency virus (HIV) and herpes virus polymerases,; this predicts that patients with CHB infection are likely to exhibit some degree of antiviral resistance to nucleoside or nucleotide monotherapies. Indeed, patients on long-term lamivudine therapy have been found to have HBV variants (YMDD variants) with reduced sensitivity to lamivudine in vitro, and have exhibited variably diminished therapeutic responses.

A fixed dose combination (FDC) formulation of lamivudine and adefovir dipivoxil for the treatment of CHB. Lamivudine (Heptodin) an active triphosphate (3TC-TP) incorporating into growing DNA chains results in premature chain termination thereby inhibiting HBV DNA synthesis. Adefovir dipivoxil (Hepsera) is an orally bioavailable pro-drug of adefovir, a nucleotide analog of adenosine monophosphate. It can inhibit both the reverse transcriptase and DNA polymerase activity and is incorporated into HBV DNA causing chain termination.

A FDC would therefore combine the established benefits of two important anti-HBV antiviral drugs, representing the first combination product for the treatment of CHB. In addition to the enhanced efficacy afforded by combination therapy, the use of a combination product could enhance convenience and compliance and ensure that patients receive the two drugs needed.

This study will evaluate the bioequivalence of a FDC containing (lamivudine 100 mg/adefovir dipivoxil 10 mg) compared to Heptodin100 mg and Hepsera 10 mg. This dose was selected as both Heptodin 100 mg and Hepsera 10 mg are approved in the PRC for the treatment of CHB. Based on extensive clinical experience with the use of both drugs either as monotherapy or in combination, it is anticipated that the co-administration of both agents in the FDC formulation will be well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician.
* Male 18 and 55 years of age.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods.
* Body weight >50 kg (110 lbs) and body mass index (BMI) between 19.0 and 25.0.
* Capable of giving written informed consent.
* QT interval corrected according to Bazzett's formula (QTcB) or QT interval corrected according to Fridericia's formula (QTcF) <450 msec; or QTc <480 msec in subjects with Bundle Branch Block.
* AST, ALT, alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening history, physical or laboratory examination, or any other medical condition or circumstance making the subject unsuitable for participation in the study.
* Treatment with any prescription or non-prescription drugs (including vitamins, herbal and dietary supplements, as well as grapefruit-containing products) within 7 days or five half-lives prior to first dose of study medication and until the end of the study. Excluded from this list is acetaminophen at doses of <=2 grams/day.
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding Day 1 of treatment period 1.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Positive urine drug screen (UDS) or breath alcohol test at screening. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Positive for hepatitis B, hepatitis C or HIV.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Electrocardiogram findings as follows (a single repeat is allowed for eligibility determination):

Parameter Males Heart rate <45 and >100 beats per minute PR Interval <120 and >220 msec QRS duration <70 and >120 msec QTc interval (Bazett) >450 msec

* Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrio-ventricular block [second degree or higher], Wolf Parkinson White syndrome).
* Sinus pauses >3 seconds.
* Any significant arrhythmia which, in the opinion of the principal Investigator and GlaxoSmithKline medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

  * Documented history of low blood pressure (BP; average systolic BP<=90 mmHg and/or diastolic BP <=45 mm Hg) or blood pressure below these values at time of screening.
  * Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
  * History of asthma or chronic obstructive pulmonary disease.
  * History of sensitivity to heparin, heparin- induced thrombocytopenia, or sensitivity to any of the study medications or components thereof.
  * History of anaphylaxis or anaphylactic reactions or severe allergic responses to drugs.
  * History of angioedema.
  * Unwillingness or inability to follow the procedures outlined in the protocol or inability to provide written informed consent.
  * Subject is mentally or legally incapacitated

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02-21 (Actual); Primary Completion 2011-04-12 (Actual); Study Completion 2011-04-12 (Actual)

PRIMARY OUTCOMES:
AUC of lamivudine | 48 hours
Cmax of lamivudine | 48 hours
AUC of adefovir dipivoxil | 48 hours
Cmax of adefovir dipivoxil | 48 hours

SECONDARY OUTCOMES:
PK parameters: t1/2 of lamivudine | 48 hours
Tolerability will be assessed by clinical data from Adverse Event reporting, nurse/physician observations, vital signs, ECGs, and clinical laboratory. | 48 hours
PK parameters: Tmax of lamivudine | 48 hours
PK parameters: Tmax of adefovir dipivoxil | 48 hours
PK parameters: t1/2 of adefovir dipivoxil | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Fok BS, Gardner S, Piscitelli S, Chen S, Chu TT, Chan JC, Tomlinson B. Pharmacokinetic properties of single-dose lamivudine/adefovir dipivoxil fixed-dose combination in healthy Chinese male volunteers. Clin Ther. 2013 Jan;35(1):68-76. doi: 10.1016/j.clinthera.2012.12.001. Epub 2012 Dec 28. PMID 23274144
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114957 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114957?search=study&study_ids=114957#rs
- Available data/document: Informed Consent Form: 114957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register